CLINICAL TRIAL: NCT06859567
Title: Proving the Efficacy of the Chester Step Test in Scleroderma Patients Compared with the 6-Minute Walk Test
Brief Title: Chester Step Test: is It Effective in Scleroderma Patients?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Havvagül Doğan, Physiotherapy and Rehabilitation, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/03-16
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Systemic Sclerosis (SSc); Chester Step Test; 6 Minutes Walk Test
Keywords: Chester step test; Systemic Sclerosis; 6 minutes walk test; Modified Borg Scale
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluated Group (Active Comparator): 6 minute walk test, Chester step test
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Comparison of the 6-minute walk test and Chester step test, one of the aerobic capacity tests

SUMMARY:
Systemic sclerosis (SSC) is a chronic autoimmune disease in which autoimmune features are associated with vascular manifestations. Patients with SSC experience many problems such as interstitial lung disease (ILD), pulmonary arterial hypertension (PAH), heart failure, severe gastrointestinal tract (GIT) involvement and scleroderma renal crisis (SRC). Because of these problems, SSC patients may develop an abnormal pulmonary hemodynamic response during exercise. In this situation, measuring the aerobic capacity of SSC patients can be a useful tool for health promotion. There are many different methods for measuring aerobic capacity tests. The most commonly used aerobic capacity test in SSC patients is the 6-minute walk test (6 MWT). However, although the 6 MWT is a commonly used test, it has some disadvantages. Because SSC affects multiple organs, there are doubts about the 6 MWT's ability to accurately assess these diseases. These disadvantages of the 6MWT have led to the search for new tests. The Chester step test (CST) is a submaximal test and a good option to assess aerobic capacity. An adapted version of the CST for non-healthy individuals can be used to assess aerobic capacity. There are some studies conducted with CST. As a result of my research, no study evaluating CST in individuals with SSC was found.

DETAILED DESCRIPTION:
Systemic sclerosis (SSC) is a chronic autoimmune disease with autoimmune features combined with vascular manifestations. Systemic sclerosis (SSC), the main symptom of which is skin sclerosis, is a marker that can detect the activity of the disease. Apart from skin involvement, SSC affects many internal organs such as the musculoskeletal system, gastrointestinal system, lungs, heart and kidneys. Because of these problems, SSC patients may develop an abnormal pulmonary hemodynamic response during exercise. This can lead to symptoms of dyspnea, fatigue and decreased exercise tolerance. In this situation, measuring the aerobic capacity of SSC patients can be a useful tool in health promotion. There are many different methods for measuring aerobic capacity tests. The most commonly used aerobic capacity test in SSC patients is the 6-minute walk test (6 MWT). However, although the 6 MWT is a commonly used test, it has some disadvantages. Because SSC affects multiple organs, there are doubts about the 6 MWT's ability to accurately assess these diseases. For an accurate 6MWT assessment, a 30 meter corridor is needed. This length of corridor is impossible to access in some clinics. These disadvantages of the 6MWT have led to the search for new tests. The Chester step test (CST) is a submaximal test and a good option for assessing aerobic capacity. Compared to 6 MWT, CST has the advantage of requiring portable equipment. It is a cost-effective option to assess exercise tolerance, fatigue and dyspnea. Because of these advantages of the CST, it can be used to assess aerobic capacity when adapted to non-healthy individuals. There are some studies conducted with CST. As a result of my research, no study evaluating CST in individuals with SSC was found. The study will be conducted at Firat University Hospital and 45 patients will be evaluated. After the demographic data of the patients included in the study are recorded, 6MWT will be performed and the results will be recorded. Then CST will be performed and the results will be recorded.6 Dyspnea, fatigue and leg fatigue will be evaluated with the Modified Borg Scale before and after MWT and CST. The patient's heart rate, oxygen saturation and blood pressure will be recorded before and after the tests. In addition, the patient's heart rate and oxygen saturation will be recorded after each level passed in CST.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Patients who can walk independently without an assistive device

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Myocardial infarction history
* Congestive heart failure
* Serious or unstable illness that may limit exercise tolerance
* Presence of severe musculoskeletal and joint disorders that may interfere with the conduct of the test
* Inability to perform the simplest level of the Chester step test
* Arthroplasty or major operations on knee and hip joints
* Uncontrolled hypertension
* Lack of ability to understand and implement all recommended procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-11 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Modified Borg Scale | up to 30 minutes
  The modified Borg scale is a validated scale for subjective perception of dyspnea used with the 6MWT to confirm the degree of respiratory distress. Exercise intensity is determined by individualized measurement. The 2002 guidelines of the American Thoracic Society recommend the modified Borg scale as an adjunct to the 6MWT. This scale is a vertical scale measured from 0 to 10. Here 0 represents no symptoms and 10 represents maximum symptoms. In this study, the modified Borg scale will be used to rate dyspnea and leg fatigue. The Borg scale will be printed out and this printout will be used for patient enumeration. The patient will be told what the numbers from 0 to 10 on the Borg scale mean. After instructions have been given, the patient will be asked to rate dyspnea and leg fatigue before and after the test and the numbers will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Merkez, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No